CLINICAL TRIAL: NCT00763412
Title: Pilot and Feasibility Study for the Treatment of Pre-diabetes in Patients With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arbelaez, Ana Maria (Individual)
Collaborators: Washington University School of Medicine (Other); National Institutes of Health (NIH) (NIH); Novo Nordisk A/S (Industry); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ana Maria Arbelaez, Assistant Professor in Pediatrics, Arbelaez, Ana Maria
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 05-1109; P60DK020579 (NIH)
Record Dates: First submitted 2008-09-29; First posted 2008-10-01 (Estimated); Results first posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Cystic Fibrosis Related Diabetes; Pancreatic Insufficiency
Keywords: Cystic Fibrosis; Diabetes; Cystic Fibrosis Related Diabetes; Pre-diabetes; oral hypoglycemic agents; Repaglinide; treatment; inflammatory markers; Lung function; nutrition
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Cystic Fibrosis; Diabetes Mellitus; Glucose Intolerance | interventions — repaglinide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1 Placebo (Placebo Comparator): 1 pill before each meal 3-4 times a day for 2 years. All subjects had abnormal glucose tolerance. Subjects were randomized to placebo or drug.
  Interventions: Drug: placebo
- 2. repaglinide (Experimental): repaglinide 0.5 mg before each meal 3-4 times a day for 2 years. All subjects had abnormal glucose tolerance.Subjects were randomized to placebo or drug.
  Interventions: Drug: repaglinide

INTERVENTIONS:
Drug: placebo — CF pancreatic insufficient patients with impaired glucose tolerance (IGT) or CFRD without fasting hyperglycemia (CFRD-No FH) by OGTT will be treated with placebo by taking 1 pill before each meal that contains more than 20 grams of carbohydrate 3-4 times a day for 2 years.
  Arms: 1 Placebo
Drug: repaglinide — CF pancreatic insufficient patients with impaired glucose tolerance (IGT) or CFRD without fasting hyperglycemia (CFRD-No FH) by OGTT will be treated with repaglinide 0.5 mg before each meal that contains more than 20 grams of carbohydrate 3-4 times a day for 2 years.
  Other Names: Prandin
  Arms: 2. repaglinide

SUMMARY:
The purpose of this study is to provide the necessary data and experience to design a larger, full scale clinical trial to determine if a certain medicine (repaglinide), which increases the amount of insulin secreted by the pancreas, can improve the nutritional status and pulmonary function of adolescents and young adults with cystic fibrosis and prediabetes by improving blood glucose control. The investigators are also trying to determine the relationship between systemic inflammatory factors and glucose impairment.

DETAILED DESCRIPTION:
As people with Cystic Fibrosis (CF) are living well into adulthood new complications are arising. CF-Related Diabetes (CFRD) has emerged as a major complication. Years prior to the diagnosis of CFRD, patients have decreasing insulin secretion, glucose intolerance, deteriorating pulmonary function, and nutritional impairment. There are no current standard recommendations for the treatment of CF patients with prediabetes, and there is little evidence that treatment of this prediabetic state in CF patients will prevent the deterioration of the lung function, nutritional status and potentially slow the progression to manifest CFRD.

To determine the feasibility of testing this hypothesis, we will perform a pilot, double-blinded, randomized controlled trial in 20 CF pancreatic insufficient patients ages of 12 to 24 years old with impaired glucose tolerance test (IGT) or CFRD without fasting hyperglycemia (CFRD-No FH) and assign them to either placebo or Repaglinide 0.5 mg PO 3 - 4 times a day before meals for two years. Patients will monitor their blood glucose daily and will be followed every 3 months for 2 years to determine changes in nutritional status by BMI and DEXA, lung function tests, frequency of hospitalizations, antibiotic courses, and degree of glucose tolerance, insulin secretion and insulin sensitivity.

In addition, based on the evidence of increased inflammation in type 2 diabetes, correlation of systemic inflammatory response at different degrees of glucose tolerance and after treatment, will be assessed in these subjects, as well as in another 20 CF pancreatic insufficient matched patients with normal glucose tolerance who will be studied once without intervention

ELIGIBILITY:
Inclusion Criteria:

* Male or females 12 -24 years old
* Diagnosis of Cystic Fibrosis by sweat test with exocrine pancreatic insufficiency
* Must have a glucose pattern by Oral Glucose Tolerance Test with fasting blood glucose <126 mg/dl and 2 hour: 140 - 199 mg/dl or >200 mg/dl.
* Weight must be stable within 5% for 3 months prior to initiation visit
* Must be able to reproducibly perform spirometry based on American Thoracic Society guidelines

Exclusion Criteria:

* Patients receiving growth hormone therapy or taking insulin
* Patients with evidence of liver dysfunction
* Patients who are status-post lung or liver transplantation
* Patients who have received systemic steroids for more than 28 days during the 6 months prior to the study
* Patients with active ABPA on steroids
* Patients taking medications that affect glucose metabolism or contraindicated with repaglinide

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2006-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil H White, M.D., Study Chair — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided
The outcome was inconclusive for this hypothesis, but the data may be valuable in future research. We are not currently sharing data from this project.

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: 1 pill before each meal 3-4 times a day for 2 years.
  placebo: CF pancreatic insufficient patients with prediabetes by OGTT will be treated with placebo by taking 1 pill before each meal that contains more than 20 grams of carbohydrate 3-4 times a day for 2 years.
- 2. Repaglinide: repaglinide 0.5 mg before each meal 3-4 times a day for 2 years.
  repaglinide: CF pancreatic insufficient patients with prediabetes by OGTT will be treated with repaglinide 0.5 mg before each meal that contains more than 20 grams of carbohydrate 3-4 times a day for 2 years.
Period: Overall Study
Arm/Group | Placebo | 2. Repaglinide
Started | 8 | 8
Completed | 4 | 4
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Population: Patients attended the Washington University CF Clinics between 2006 and 2008.
Groups:
- Patients Who Received Placebo; Patients Who Received Repaglinide: All participants were receiving ADEK vitamins and pancreatic enzyme replacement. Patients were required to be clinically stable, without evidence of deterioration from previous pulmonary function tests (PFTs) for 3-months prior to the study and without CF exacerbation or hospitalization for 2-months prior to the study. Additionally, patients were required to have maintained stable weight within 5% variance for 3-months prior to participation. Exclusion criteria included fasting blood glucose levels >126 mg/dL on study day, IV antibiotic or systemic steroid use within two months, oral corticosteroid usage for more than 28-days over the past 6-months, history of lung or liver transplant, elevated transaminases, allergic bronchopulmonary aspergillosis, or the inability to perform spirometry.
- Total: Total of all reporting groups
Arm/Group | Patients Who Received Placebo | Patients Who Received Repaglinide | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants] — Patients attended the Washington University CF Clinics between 2006 and 2008.
  Participants
    <=18 years | 3 | 3 | 6
    Between 18 and 65 years | 1 | 1 | 2
    >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 16 [12 to 18] | 15 [12 to 22] | 15.5 [12 to 22]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16
BMI [Mean (Full Range); unit: Kg/m^2] | 19.45 [14.55 to 22.96] | 18.38 [16.78 to 20.3] | 18.94 [14.55 to 22.96]
Wt Z score [Mean (Full Range); unit: Z score] | -1.11 [-1.84 to 0.33] | -0.29 [-0.75 to 0.19] | -0.7 [-1.84 to .33]
Fat % [Mean (Full Range); unit: % Fat mass] | 20.34 [7.36 to 38.74] | 22.06 [9.76 to 28.81] | 21.2 [7.36 to 38.74]
Lean % [Mean (Full Range); unit: % Lean mass] | 76.71 [58.6 to 89.67] | 75 [68.22 to 87.11] | 75.9 [58.6 to 89.67]
Tanner stage [Mean (Full Range); unit: units on a scale] — This is a measurement of puberty development. This is a 1-5 scale describing 1 as the least developed and 5 as the most developed in puberty.
  units on a scale | 3.75 [2 to 5] | 3.25 [1 to 5] | 3.5 [1 to 5]
FEV 1 [Mean (Full Range); unit: % of lung function] | 97.75 [92 to 121] | 92.75 [70 to 105] | 95.25 [70 to 121]
Fasting Glucose [Mean (Full Range); unit: mg/dl] — This was the baseline glucose in a 2 hour oral glucose tolerance test. (OGTT)
  mg/dl | 99.1 [87 to 114.5] | 100 [94 to 106] | 99.6 [87 to 114.5]
2 hour glucose [Mean (Full Range); unit: mg/dl] — Final glucose sample in a 2 hour OGTT.
  mg/dl | 182.4 [144 to 218.5] | 183 [140 to 206] | 182.7 [140 to 218.5]
Fasting C-Peptide [Mean (Full Range); unit: mg/dl] | 1.2 [0.6 to 2.1] | 1.7 [1.0 to 3] | 1.45 [0.6 to 3]
2 hour c-peptide [Mean (Full Range); unit: mg/dl] — final c-peptide measurement at the end of 2 hour OGTT.
  mg/dl | 9.7 [6 to 15.5] | 9.5 [5 to 12.6] | 9.6 [5 to 15.5]
Inflammatory marker [Mean (Full Range); unit: pg/ml] — baseline values collected during a 2 hour OGTT.
  pg/ml
    IL1 | 0.1 [0.1 to 1.9] | 0.9 [.01 to 1.7] | 0.5 [0.1 to 1.9]
    IL6 | 8.3 [1.5 to 26.4] | 12.6 [3.7 to 33.8] | 10.5 [1.5 to 33.8]
    IL8 | 7 [2.7 to 17.8] | 8.5 [4.6 to 13.6] | 7.75 [2.7 to 17.8]
    TNF Alpha | 7.3 [5.2 to 7.3] | 4.5 [2.5 to 6.4] | 5.9 [2.5 to 7.3]
CRP [Mean (Full Range); unit: mg/L] — inflammatory marker
  mg/L | 1.8 [0.2 to 2.5] | 2.1 [0.8 to 3.3] | 1.95 [0.2 to 3.3]

OUTCOME MEASURES:

1. Primary Outcome: BMI
Time Frame: 2 year/end of study
Measure: Mean (Full Range); unit: Kg/m^2
Groups:
- 1 Placebo: 1 pill before each meal 3-4 times a day for 2 years.
  placebo: CF pancreatic insufficient patients with prediabetes by OGTT will be treated with placebo by taking 1 pill before each meal that contains more than 20 grams of carbohydrate 3-4 times a day for 2 years.
Arm/Group | 1 Placebo | 2. Repaglinide
Number analyzed (Participants) | 4 | 4
Kg/m^2 | 19.63 [15.56 to 22.64] | 21.19 [20.78 to 21.8]

2. Primary Outcome: Body Composition
Description: Reporting % of Fat and Lean body mass
Time Frame: 2 year/end of study
Measure: Mean (Full Range); unit: % body mass
Arm/Group | 1 Placebo | 2. Repaglinide
Number analyzed (Participants) | 4 | 4
% body mass
  Fat | 19.82 [12 to 37.8] | 26.21 [8.78 to 34.26]
  Lean | 77.15 [59.54 to 87.84] | 70.83 [62.82 to 87.8]

3. Primary Outcome: CRP
Time Frame: 2 year/end of study
Measure: Mean (Full Range); unit: mg/L
Arm/Group | 1 Placebo | 2. Repaglinide
Number analyzed (Participants) | 4 | 4
mg/L | 9.6 [0.7 to 27.5] | 2 [0.6 to 3.7]

4. Secondary Outcome: Glucose Tolerance
Description: We completed the OGTT at the 2 year/end of study visit.
Time Frame: 2-year
Measure: Mean (Full Range); unit: mg/dl
Arm/Group | 1 Placebo | 2. Repaglinide
Number analyzed (Participants) | 4 | 4
mg/dl
  fasting glucose | 101.5 [91 to 121] | 94.5 [85 to 108]
  2 hour glucose | 185.75 [145 to 258] | 184 [123 to 266]

5. Secondary Outcome: Inflammatory Markers
Time Frame: 2 year/end of study
Measure: Mean (Full Range); unit: pg/ml
Arm/Group | 1 Placebo | 2. Repaglinide
Number analyzed (Participants) | 4 | 4
pg/ml
  IL1 | 0.14 [0.13 to 0.17] | 0.34 [0.13 to 1]
  IL6 | 10.4 [0.54 to 28.6] | 6 [2.2 to 11.9]
  IL8 | 5.8 [3.59 to 10.79] | 5.2 [3.1 to 8.33]
  TNF alpha | 5.1 [2.05 to 7.5] | 3.6 [1.99 to 5.3]

6. Secondary Outcome: Wt Z Score
Time Frame: 2 year/end of study
Measure: Mean (Full Range); unit: Z score
Arm/Group | 1 Placebo | 2. Repaglinide
Number analyzed (Participants) | 4 | 4
Z score | -1.21 [-1.94 to 0.08] | -0.26 [-0.31 to 0.72]

7. Secondary Outcome: Tanner Stage
Description: Puberty scale measuring 1-5, 1 being least development, 5 being most development.
Time Frame: 2 year/end of study
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | 1 Placebo | 2. Repaglinide
Number analyzed (Participants) | 4 | 4
units on a scale | 4.25 [4 to 5] | 5 [5 to 5]

8. Secondary Outcome: FEV 1
Description: % of lung function
Time Frame: 2 year/end of study
Measure: Mean (Full Range); unit: % lung function
Arm/Group | 1 Placebo | 2. Repaglinide
Number analyzed (Participants) | 4 | 4
% lung function | 90.5 [71 to 99] | 91.5 [74 to 108]

9. Secondary Outcome: C-Peptide
Time Frame: 2 year
Measure: Mean (Full Range); unit: pg/ml
Arm/Group | 1 Placebo | 2. Repaglinide
Number analyzed (Participants) | 4 | 4
pg/ml
  fasting | 1.5 [0.8 to 2.3] | 1.6 [0.6 to 2.5]
  2 hour | 7.5 [5 to 8.7] | 7.7 [4.2 to 11.9]

ADVERSE EVENTS:
Time Frame: This pilot study was designed to collect data over a 2 year time period.
Description: Glucose diaries, and food diaries were reviewed, and safety labs were collected at each visit. Physical assessments by the PI were completed as well.
Groups:
- Placebo: Placebo group of CF pancreatic insufficient patients ages 12-24 years old with impaired glucose tolerance test (IGT) or CFRD without fasting hyperglycemia (CFRD-No FH).
- Repaglinide: Repaglinide intervention group of CF pancreatic insufficient patients ages 12-24 years old with impaired glucose tolerance test (IGT) or CFRD without fasting hyperglycemia (CFRD-No FH).
Arm/Group | Placebo | Repaglinide
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
A limitation of the study was the very small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No